CLINICAL TRIAL: NCT06440096
Title: Harran University Hospital Department of Physical Medicine and Rehabilitation
Brief Title: Complete Blood Count-derived Indexes in Inflammatory Modic Changes
Status: Completed | Type: Observational
Sponsor: Veysel Delen, MD (Other)
Responsible Party: Sponsor-Investigator, Veysel Delen, MD, Harran University Hospital, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Organization: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Other Study IDs: YÖMAVD
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Modic Changes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modic changes type I: 24 patients with type I Modic changes
  Interventions: Diagnostic Test: hemogram
- Modic changes type II: 24 patients with type II Modic changes
  Interventions: Diagnostic Test: hemogram

INTERVENTIONS:
Diagnostic Test: hemogram — hemogram

SUMMARY:
Some indicators generated from hemogram such as neutrophil/lymphocyte (NLR) have been suggested as biomarkers of systemic inflammation. Type I Modic changes (MCs) have inflammatory nature histologically and are more painful clinically than type II MCs. Therefore, we hypothesized that patients with type I MCs may have increased inflammatory biomarkers and low back pain than those with type II MCs. The aim of this study was to test this hypothesis.

DETAILED DESCRIPTION:
Patients and Methods: A total of 48 patients with MCs (type I/type II=24/24) were included in this study. Their demographic, clinical and hematologic characteristics were recorded. A 10 cm Visual Analog Scale (VAS) was used to detect low back pain intensity. Systemic inflammatory biomarkers including NLR, monocyte/lymphocyte (MLR), platelet/lymphocyte (PLR), neutrophil/lymphocyte*platelet (NLPR), systemic inflammatory index (SII), systemic inflammatory response index (SIRI), and aggregate index of systemic inflammation (AISI) were derived from whole blood cell count.

Keywords: Neutrophil-to-lymphocyte ratio, inflammation, Modic changes, back pain.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were male or female with type I or type II MCs, aged ≥18 and ≤64 years old, and accepted informed consent to participation.

Exclusion Criteria:

* type III MCs and a combination of MCs' types were excluded. In addition, acute low back pain, spinal deformities, inflammatory diseases, cancers, heart diseases, stroke, lactation, pregnancy, psychiatric disorders, and extreme obesity (BMI≥40 kg/m²) were also excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male or female patients with type I or type II Modic changes, aged ≥18 and ≤64 years old
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Hemogram-derived inflammation indexes | 10 minutes
  blood-based

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Şanlıurfa, Sanliurfa, Turkey (Türkiye)